CLINICAL TRIAL: NCT06552013
Title: Action Towards Health Equity and Improved Air Quality in the Duwamish Valley: A Multilevel Asthma Intervention
Acronym: DAISY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Anjum Hajat, Associate Professor: School of Public Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00018735; 1R01ES034749-01 (NIH)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Asthma in Children
Keywords: air quality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham filter (Experimental): Participants in this arm will receive a sham filter for their box fans. These filters receive a MERV rating of 1 and only filter very large particles and debris such as lint, hair and insects. These particles have little to no impact on asthma symptoms. MERV stands for "minimum efficiency reporting value" and a filter receives a MERV rating as determined by the American Society of Heating, Refrigeration, and Air-Conditioning Engineers.
  Interventions: Other: Sham filter
- MERV 13 filter (Experimental): Participants in this arm will receive a MERV 13 filter for their box fans. MERV 13 filters trap the majority of small particles, as small as 1 micron. It also traps up to 75% of particles that are as small as 0.3 microns.
  Interventions: Other: MERV 13 filter

INTERVENTIONS:
Other: MERV 13 filter — This is an environmental intervention consisting of a low-cost box fan with a MERV 13 filter placed behind it. The company Lasko makes these fans and other environmental appliances.
  Arms: MERV 13 filter
Other: Sham filter — This is an environmental intervention consisting of a low-cost box fan with a sham filter (MERV 1) placed behind it. The company Lasko makes these fans and other environmental appliances.
  Arms: Sham filter

SUMMARY:
The goal of this randomized control trial is to learn if box fans and filters can reduce asthma symptoms and improve indoor air quality in children ages 6 - 17 years old with asthma living in the Duwamish Valley, Seattle, Washington. The main question it aims to answer are:

* Do box fans with filters improve asthma symptoms?
* Do box fans with filters improve an objective measure used to monitor lung function known as forced expiratory volume during the first second (FEV1)? Researchers will compare children living in households with high quality filters to those in households with sham filters to see if air quality and asthma symptoms improve.

Participants will

* fill out several questionnaires
* monitor their lung function with a peak flow meter
* place an air monitor in their homes to monitor indoor air quality
* run the box fan when they are at home

ELIGIBILITY:
Inclusion Criteria:

* age (6-17 years)
* poorly controlled physician diagnosed asthma defined as more than four days with asthma symptoms in the past two weeks, use of asthma rescue medication for more than four days in the past two weeks, or health care utilization due to asthma in the past year (hospitalization, emergency room visit, or unscheduled clinic visit)
* living in Georgetown and South Park neighborhoods of Seattle

Exclusion Criteria:

* children with unstable housing or shared custody arrangements

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Asthma symptoms | ACQ will be measured weekly for 6 consecutive weeks, two pre-intervention weeks (before box fans have been given to participant) and four weeks while fans are being used in the home. Symptoms will also be assessed at the six month follow-up visit.
  Symptoms are evaluated with the seven-item asthma control questionnaire (ACQ), a validated tool used in children.
FEV1 | FEV1 measures will be taken daily, once in the morning and once at night for the six week study time frame. Prior to the six month follow up we will ask participants to take three consecutive days of FEV1 measurements, for an additional 6 measures
  FEV1 is captured with a digital peak flow meter.

SECONDARY OUTCOMES:
Asthma quality of life | Will be evaluated at baseline (visit 1), after 6 weeks (visit 3) and at 6 month follow up (visit 4)
  Will be assessed with the15-item mini-asthma quality of life questionnaire, a validated tool
Use of rescue medications | ACQ will be measured weekly for 6 consecutive weeks, two pre-intervention weeks (before box fans have been given to participant) and four weeks while fans are being used in the home. Symptoms will also be assessed at the six month follow-up visit.
  This is an item on the ACQ. See primary outcome.
Health care utilization in the past month | Will be evaluated at baseline (visit 1), after 6 weeks (visit 3) and at 6 month follow up (visit 4)
  Will be assessed with the six-item asthma-related health care utilization questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anjum Hajat, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Duwamish River Community Coaltion, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual level data sets will be shared. Given the small sample size of our study, we will protect against deductive disclosure by withholding information that could result in disclosure.
  We will also require interested investigators to provide a proposal that will outline their study question and analytic methods. If there is any overlap with ongoing manuscripts, we will ask investigators to collaborate with ongoing efforts or to propose an alternative study question. Investigators will be required to sign a data sharing agreement that will include assurances about participant privacy and data confidentiality.
  We do not anticipate a great number of requests for our data so will handle them on an individual basis. After discussing the data with investigators who are interested in accessing it, we will share it via a secure site.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Health data from our randomized control trial will be shared with interested investigators after the two main results papers from the study have been accepted for publication (one on asthma outcomes and the other on air quality). Since data collection will not be finished until year four of the study and the analysis and writing will take some time, data sharing will likely occur after the grant period has ended.